CLINICAL TRIAL: NCT06130527
Title: Comparison of the Effects of Nicardipine and Remifentanil on Surgical Visual Field and Hemodynamic Parameters in Tympanomastoidectomy Cases
Brief Title: Comparison of the Effects of Nicardipine and Remifentanil on Surgical Visual Field
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erol Karaaslan (Other)
Responsible Party: Sponsor-Investigator, Erol Karaaslan, Associate Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: erolkaraaslan5
Record Dates: First submitted 2023-09-15; First posted 2023-11-14 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Other Complications of Surgical and Medical Procedures
Keywords: Surgical visual field; nicardipine; remifentanil
MeSH Terms: interventions — Nicardipine; Remifentanil

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective Randomized, Placebo-Controlled Clinical Tria
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicardipine (Active Comparator): Nicardipine is a dihydropyridine derivative vasoselective drug. Rapid onset of action i.v. nicardipine is used when rapid control of blood pressure is needed. The potential role of i.v. nicardipine was shown in many cardiovascular and neurovascular surgical procedures and surgical procedures in which CH was performed with hemostasis (6).
  Interventions: Procedure: Nicardipine
- Remifentanil (Active Comparator): Although remifentanil has unique pharmacokinetic properties, its pharmacodynamic effects are similar to those of other opioids. Remifentanil has dose-dependent analgesic, sedation and respiratory suppression side effects. All of these effects are antagonized by the mu receptor-specific opioid antagonist naloxone. Remifentanil has vagotonic and sympatholytic effects, and common side effects are bradycardia (heart rate <50 beats/min) and hypotension (SBP <80 mm Hg). Other common side effects are itching, nausea and vomiting, and chest wall stiffness after bolus administration (35).
  The elderly population is more sensitive to opioid effects. It has been shown that it suppresses the delta wave in EEG due to the effects of opioids in the cerebral cortex. This feature is twice as common in the elderly as in the younger population.
  Interventions: Procedure: Remifentanil

INTERVENTIONS:
Procedure: Nicardipine — Following the intubation, the infusion was initiated by using an infusion device (Orchestra Base Primea, Fresenius Kabi) with an i.v. dose of 1.0 µg/kg/min iv in Group N. The targeted MAP was determined as 50-65 mmHg and drug doses were increased until the targeted MAP was achieved In Group N. Nicardipine infusion will be increased by titration in groups with MAP above 65 mm/Hg for more than 5 minutes.
  Arms: Nicardipine
Procedure: Remifentanil — Infusion was administered i.v. using an infusion device (Orchestra Base Primea, Fresenius Kabi). In Group R, the dose will start at 0.05 µg/kg/min following intubation. The target MAP was determined as 50-65 mmHg and drug doses will be increased until the target MAP is reached. HR more than 120 seconds and less than 45 beats/min will be considered as bradycardia and the remifentanil dose will be reduced. If response is unsatisfactory, 0.5 mg Atropine i.v. will be implemented. Nicardipine and Remifentanil infusions in groups will be increased by titration if MAP rises above 65 mm/Hg for more than 5 minutes.
  Arms: Remifentanil

SUMMARY:
In the present study, the purpose was to compare the effects of Nicardipine and Remifentanil on surgical visual field and hemodynamic parameters in microscopic tympanomastoidectomy cases with Controlled Hypotension (CH).

DETAILED DESCRIPTION:
The visibility of the surgical field provides many advantages (e.g., preventing possible complications and reducing the duration of surgical application). In microsurgery performed in a closed and narrow area (e.g., middle ear surgery), even a small amount of blood may impair the quality of vision in the operation area and complicate the surgical intervention.

Controlled Hypotension (CH) is often preferred in some planned surgeries in reducing intraoperative bleeding, creating a quality surgical field, increasing surgical success, and reducing surgical complications. It is especially important to use it in interventions such as Functional Endoscopic Sinus Surgery (FESS), septoplasty, tympanoplasty, and vertebral surgery performed with microsurgery. As well as the advantages of CH, there is the possibility of causing various side effects by causing target organ hypoperfusion. Cerebral, renal, liver, and cardiovascular systems are the organs most affected by side effects.

Various hypotensive agents such as volatile anesthetics, sympathetic antagonists, sodium nitroprusside, nitroglycerin, hydralazine, trimethaphan, and α2 agonists are used in the literature to provide controlled hypotension.

Nicardipine is a dihydropyridine derivative vasoselective drug. Rapid onset of action i.v. nicardipine is used when rapid control of blood pressure is needed. The potential role of i.v. nicardipine was shown in many cardiovascular and neurovascular surgical procedures and surgical procedures in which CH was performed with hemostasis.

Its dromotropic effect is very low because nicardipine has no significant depressant effect on the conduction system and electrophysiological parameters of the heart. It undergoes substantial presystemic elimination in the liver after oral administration. For this reason, the rate of elimination does not change in patients with kidney failure. The elimination half-life is approximately 2 hours and slows down in patients with hepatic dysfunction.

Many studies investigate the effects of CH on surgical field image quality, surgical satisfaction, bleeding, and hemodynamic parameters. However, in our literature review, no study was detected comparing Nicardipine and Remifentanil in microscopic tympanomastoidectomy cases.

In the present study, the purpose was to compare the effects of controlled hypotension with nicardipine and remifentanil on the quality of surgical field visibility and hemodynamic parameters in endoscopic tympanomastoidectomy cases

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients of both sexes,
* aged 18-65 years,
* scheduled for tympanomastoidectomy and decided to perform CH,

Exclusion Criteria:

* hypertension,
* anticoagulant medication,
* pregnancy
* major hepatic,
* renal,
* cerebral, or cardiorespiratory dysfunction,
* neurological or psychiatric disease
* ASA 3-4,
* Body Mass Index BMI≥35 kg/m2,
* difficult intubation was considered (Mallampati score 3-4, a thyromental distance less than 6 cm, maximum mouth opening less than 3 cm),
* the number of intubation attempts more than two, cases with allergies to any of the agents used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of the intraoperative surgical field | Measurements will be made at four different times B1: Skin incision (initial stage of surgery), B2: mastodectomy stage of surgical intervention, B3: cholestatum cleaning stage of surgical intervention, B4: grafting phase of surgical intervention
  Quality of the intraoperative surgical field will be measured on a grade of 0-10 (0-1. no bleeding, 2-3. mild bleeding, 4-5. Mild to moderate bleeding, 6-7. moderate bleeding, 8-9. moderate to severe bleeding, 10. Severe bleeding)

SECONDARY OUTCOMES:
Heart rate | Measurements will be made at six different times T1: at the 20th minute of surgical intervention T2: mastodectomy stage of intervention T3: cholestatum clearing of intervention T4: grafting phase of surgical T5: first minute after extubation, T6: 10 min
  Heart rate is measured as beats/minute on the anesthesia monitor
Mean arterial pressure | Measurements will be made at six different times T1: at the 20th minute of surgical intervention T2: mastodectomy stage of intervention T3: cholestatum clearing of intervention T4: grafting phase of surgical T5: first minute after extubation, T6: 10 min
  Mean arterial pressure is measured as mmHg on the anesthesia monitör

CONTACTS AND LOCATIONS:
Overall Officials: Erol Karaaslan, assoc prof, Study Director — Inonu University Medical Faculty , malatya.turkey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker AR, Baker AB. Anaesthesia for endoscopic sinus surgery. Acta Anaesthesiol Scand. 2010 Aug;54(7):795-803. doi: 10.1111/j.1399-6576.2010.02259.x. Epub 2010 Jun 16. PMID 20560885
- [Result] Shin S, Lee JW, Kim SH, Jung YS, Oh YJ. Heart rate variability dynamics during controlled hypotension with nicardipine, remifentanil and dexmedetomidine. Acta Anaesthesiol Scand. 2014 Feb;58(2):168-76. doi: 10.1111/aas.12233. Epub 2013 Nov 22. PMID 24261345